CLINICAL TRIAL: NCT05676034
Title: A Phase II Study of Safety and Efficacy of AMX0035 in Adult Patients With Wolfram Syndrome
Brief Title: AMX0035 in Adult Patients With Wolfram Syndrome
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amylyx Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A35-008
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Wolfram Syndrome
Keywords: Wolfram; Wolfram syndrome
MeSH Terms: conditions — Wolfram Syndrome | interventions — sodium phenylbutyrate and taurursodiol; 4-phenylbutyric acid

STUDY DESIGN:
Intervention Model Description: A 144 week open-label treatment period of AMX0035 administered twice daily
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMX0035 (Experimental): AMX0035 administered by mouth for 144 weeks: Once daily for first 3 weeks and then twice daily for the remainder of the study if tolerated by participant
  Interventions: Drug: AMX0035

INTERVENTIONS:
Drug: AMX0035 — AMX0035
  Other Names: Proprietary formulation of taurursodiol and sodium phenylbutyrate

SUMMARY:
This study is an open label Phase II study to evaluate the safety and efficacy of AMX0035 in adults with Wolfram syndrome.

DETAILED DESCRIPTION:
AMX0035 is a combination therapy designed to reduce neuronal death through blockade of key cellular death pathways originating in the mitochondria and endoplasmic reticulum (ER). This clinical trial is designed to demonstrate that treatment is safe, tolerable, and to evaluate the effect of AMX0035 on residual beta cell functions by monitoring c-peptide levels during a 0-240 minute mixed-meal tolerance test. The trial will also assess the effects of AMX0035 on changes to diabetic measurements including daily insulin dose, time in good glucose range, and HbA1c levels. Effect on best-corrected visual acuity in both eyes will also be evaluated.

ELIGIBILITY:
Key Inclusion Criteria:

* Definitive diagnosis of Wolfram syndrome
* Insulin dependent diabetes mellitus due to Wolfram syndrome
* At least 17 years of age
* Participant must be willing to wear a CGM device for the duration of the study

Key Exclusion Criteria:

* Presence of pathologies that can alter the enterohepatic circulation of bile acids (e.g., ileal resection and stoma, regional ileitis)
* Any history of heart failure per New York Heart Association (NYHA)
* History of or family history of breast and/or ovarian cancer
* Participant under severe salt restriction where the added salt intake due to treatment would put the patient at risk, in the Investigator's judgment
* Received treatment with any investigational drug or device within the 30 days (or 5 half-lives, whichever is longer) prior to first dose at Day 1
* Previous treatment with gene or cellular therapy

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of AMX0035 on residual beta-cell function by monitoring C-peptide levels during a 0-240 minutes mixed-meal tolerance test (MMTT) | 24 weeks
  * C-peptide area under the curve (AUC) response at Week 24 using a 0-240 minute MMTT
  * Change from Baseline in area under the curve (AUC) in delta C-peptide at Week 24 using a 0-240 minute MMTT
To assess the safety and tolerability of AMX0035 administered orally for up to 144 weeks in adult participants with Wolfram syndrome | 148 weeks
  * Incidence and severity of Adverse Events and Serious Adverse Events
  * Incidence of abnormalities in clinical laboratory assessments

SECONDARY OUTCOMES:
To evaluate the effect of AMX0035 during a 0-240 minute MMTT | 48 weeks
  C-peptide AUC response to a 240-minute MMTT at Week 48
To assess the effect of AMX0035 on visual acuity | 48 weeks
  Change from Baseline on best-corrected visual acuity for both eyes measured on the LogMAR scale by sight tests using Snellen chart at Week 48
To evaluate the effect of AMX0035 on total daily insulin dose | 24 weeks
  Change from Baseline of exogenous insulin dose to Week 24
To evaluate the effect of AMX0035 on glucose range | 24 weeks
  Change from Baseline to Week 24
  * Time in good range
  * Time below range
  * Time above range
To evaluate the effect of AMX0035 on HbA1c levels | 24 weeks and 48 weeks
  Change from Baseline to Week 24 and Week 48 in HbA1c level

CONTACTS AND LOCATIONS:
Overall Officials: Camille Bedrosian, MD, Study Director — Amylyx Pharmaceuticals
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes